CLINICAL TRIAL: NCT01521169
Title: Clinical Study for Evaluating the Plasma Cholesterol-reducing Activity of a Plant Sterol-enriched Yoghurt Drink - Effectiveness and Long-term Safety Study
Brief Title: Long-term Effectiveness Study on Cholesterol-reducing Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danone Japan (Industry)
Responsible Party: Sponsor
Organization: Danone Global Research & Innovation Center (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: NU332
Record Dates: First submitted 2012-01-26; First posted 2012-01-30 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Normal and Mild Hypercholesterolemic Subjects
Keywords: Plant sterol - Hypercholesterolemia - Diet - Dairy
MeSH Terms: interventions — Phytosterols

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- 1 = Tested product dose 1 (Active Comparator)
  Interventions: Other: 1 - low-fat dairy fermented product (drinkable) enriched with plant sterols (0,8g /day equivalent as free sterols).
- 2 = Tested product dose 2 (Active Comparator)
  Interventions: Other: 2 - low-fat dairy fermented product (drinkable) enriched with plant sterols (1,6g /day equivalent as free sterols).
- 3 = Control product (Sham Comparator)
  Interventions: Other: 3 - low-fat dairy fermented product (drinkable) without plant sterols.

INTERVENTIONS:
Other: 1 - low-fat dairy fermented product (drinkable) enriched with plant sterols (0,8g /day equivalent as free sterols). — 1 = Intervention with test product 1 (0,8g of plant sterol/day)
  Arms: 1 = Tested product dose 1
Other: 2 - low-fat dairy fermented product (drinkable) enriched with plant sterols (1,6g /day equivalent as free sterols). — 2 = Intervention with test product 2 (1,6g of plant sterol/day)
  Arms: 2 = Tested product dose 2
Other: 3 - low-fat dairy fermented product (drinkable) without plant sterols. — 3 = Intervention 3 (1 control product/day)
  Arms: 3 = Control product

SUMMARY:
The purpose of this study is to investigate the effect of consumption of a drinkable low fat fermented milk enriched with 0,8g or 1,6g of plant sterols on reducing plasma cholesterol (LDL-cholesterol) concentration during 12 weeks of product consumption.

ELIGIBILITY:
Inclusion Criteria:

1. Subject with total cholesterol plasma level between 200 mg/dL to 240 mg/dL; and LDL-cholesterol between 120 mg/dL to 160 mg/dL.
2. Subject aged from 20 to 65 years (bounds included)
3. Subject with BMI between 19 - 30 kg/m² (bounds included)
4. Subject with triglycerides under 400 mg/dL (4.6 mmol/L)
5. Non diabetic subjects (BS≤125 mg/dL)
6. Non hypertensive subjects (SBP<140mmHg and DBP<90 mmHg)
7. Subject accepting to follow the dietary recommendations advisable for hypercholesterolemic
8. Subject agreeing not to consume any other plant sterol supplements or excess plant sterol during the study period
9. Subject, upon briefing of the content of the present study, fully understanding and agreeing to its objective; and being able to personally sign a written informed consent and subject having signed the written consent to take part in the study

Exclusion Criteria:

1. Subject currently involved in a clinical trial.
2. Subject taking any dislipademia treatment (statins,ezetimibe, niacin, omega-3 FA, fibrates)
3. Subject having blood sample of 200 ml or more taken (e.g., donated blood) within 1 month, or 400 ml or more within 3 months of the start of the present study.
4. For female subject: pregnancy or intention to be pregnant during the study.
5. For female subject: breast feeding.
6. Subject presenting known allergy or history of hypersensitivity to plant sterols or dairy products.
7. Subject having lactose intolerance.
8. Subjects having sitosterolemia
9. Diabetic subject (Type I and type II)
10. Subject with heavy alcohol intake (>60g/day)
11. Subject receiving systemic treatment or topical treatment likely to interfere with evaluation of the study parameters
12. Subject receiving a transplant or under immunosuppressor treatment
13. Subject receiving treatment for serious liver, renal, cardio-vascular, respiratory, endocrine, or metabolic disorders.
14. Subject having cardiovascular history or cardiovascular events (e.g.myocardial infarction, angina pectoris, surgical or endocoronary intervention, stroke, inferior member arteriopathy, etc.) during the last 6 months
15. Subject deemed unsuitable by the investigator.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 138 (Actual)
Dates: Start 2010-02; Primary Completion 2010-07 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Senrichuo Ekimae Clinic - Senri Life Science Center 13F, Osaka, Japan